CLINICAL TRIAL: NCT04566627
Title: Acceptability and Feasibility Study of the Program "Yo Se Lo Que Quiero" (Unplugged) Aiming to Reduce Substance Use Among Adolescents in Chile: a Pilot Randomized Controlled Study.
Brief Title: Acceptability and Feasibility Study of the Program "Yo Se Lo Que Quiero" (Unplugged)
Acronym: YSLQQ-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Jorge Gaete, Associate Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Fondecyt Regular 1181724 Pilot
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Substance Use; Adolescent Behavior
MeSH Terms: conditions — Substance-Related Disorders; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: Evaluators were blinded to the intervention condition of the schools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YSLQQ group (Experimental): Schools in this group implemented "Yo Sé Lo Que Quiero" program. This is the cultural adaptation of the Unplugged program. This is a preventive intervention to reduce tobacco, alcohol, and marihuana use among adolescents. It consists of 12 sessions, delivered by a trained facilitator on a weekly basis.
  Interventions: Behavioral: "Yo Sé Lo Que Quiero" programl
- Control Group (No Intervention): Schools in this group implemented the usual preventive actions to reduce substance use. Usually, these actions are not manualized.

INTERVENTIONS:
Behavioral: "Yo Sé Lo Que Quiero" programl — "Yo Sé Lo Que Quiero" program is the cultural adaptation of the Unplugged program. This is a preventive intervention to reduce tobacco, alcohol, and marihuana use among adolescents. It consists of 12 sessions, delivered by a trained facilitator on a weekly basis.
  Other Names: Unplugged; Todojunto
  Arms: YSLQQ group

SUMMARY:
Substance use and drug related disorders are important public health problems. Alcohol and illicit drug use account for 5.4% of the total burden of disease and the peak has been found in early adulthood (between ages 20 and 30 years). Substance use is one of the leading problems among Chilean adolescents. One out of four 8 th to 12 th graders have smoked cigarettes in the last month. A 35.6% of students (37%, girls; 34.2%, boys) between Year 8 and Year 12 have reported any alcohol use during the last month. It is worrying that a third of 14 years old students report using alcohol in the last month in Chile. Furthermore, two out of three who are using alcohol, report regularly using 5 or more drinks in a row during the last month. Cannabis use among young Chileans has increased in recent years. Today, one out of five students between Year 8 and Year 12 referred cannabis use during the last 30 days. Almost a 20% of students in Year 8 have used cannabis in the last year.

Therefore, is urgent to provide evidence-based drug preventive interventions to the Chilean population, specifically to school students, to tackle this problem and reduce the risk for a more dramatic future health scenario.

The aim of this study was to assess the acceptability and feasibility of the cultural adaptation of "Yo Sé Lo Que Quiero" program. This is a pilot randomized controlled trial. The participants of this pilot were students attending six low-income primary schools in Santiago, Chile.

DETAILED DESCRIPTION:
Substance use and drug related disorders are important public health problems. Alcohol and illicit drug use account for 5.4% of the total burden of disease and the peak has been found in early adulthood (between ages 20 and 30 years). Substance use is one of the leading problems among Chilean adolescents. One out of four 8 th to 12 th graders have smoked cigarettes in the last month. A 35.6% of students (37%, girls; 34.2%, boys) between Year 8 and Year 12 have reported any alcohol use during the last month. It is worrying that a third of 14 years old students report using alcohol in the last month in Chile. Furthermore, two out of three who are using alcohol, report regularly using 5 or more drinks in a row during the last month. Cannabis use among young Chileans has increased in recent years. Today, one out of five students between Year 8 and Year 12 referred cannabis use during the last 30 days. Almost a 20% of students in Year 8 have used cannabis in the last year.

Therefore, is urgent to provide evidence-based drug preventive interventions to the Chilean population, specifically to school students, to tackle this problem and reduce the risk for a more dramatic future health scenario.

The aim of this study was to assess the acceptability and feasibility of the cultural adaptation of "Yo Sé Lo Que Quiero" program. This is a pilot randomized controlled trial. The participants of this pilot were students attending six low-income primary schools in Santiago, Chile.

This pilot study is part of a larger research project with the final aim of testing the effectiveness of "Yo Sé Lo Que Quiero" program to reduce substance use among adolescents in Chile.

ELIGIBILITY:
Inclusion Criteria for schools:

* Mixed schools (boys and girls)
* Schools with a high vulnerability index, IVESINAE > 70%. The IVESINAE is an indicator of the proportion of the students who have several risk factors regarding family income, parental education among other factors. This index is built by the Ministry of Education in Chile and help to direct resources to the schools.
* Located in the Metropolitan region in Chile.

Exclusion Criteria for schools:

* Having a structure and manualized substance use preventive program in place.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1214 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of the program by students | Inmediately Post-intervention
  A questionnaire exploring the acceptability of the program was answered by the students who participated in the intervention. This questionnaire asked about the students´opinions about the content of the intervention, strategies used, materials, and performance of the facilitators. The questionnaire also asked about satisfaction and the helpfulness of the program to improve emotions management, school climate, relationships with other people, and learning about drugs´ risks. Finally, the questionnaire asked about sense of self-efficacy to avoid drugs today and in the future.
Feasibility of the program | 1 year
  A register was used to determine the number of schools initially contacted and the number of schools that accepted to participate; number of students that consented and assented to participate in the study at baseline and at follow-up; the number of sessions planned and actually delivered; the number of schools and teachers that participated in the training.

SECONDARY OUTCOMES:
EU-Dap | One month
  The European Drug Addiction Prevention Trial Questionnaire (EU-Dap) was the instrument used to evaluate the Unplugged drug prevention program among adolescents in The European Drug Addiction Prevention (EU-Dap) trial project which took place between 2003-2005. EU-Dap was granted by the European Commission within the 2002 and 2005 Public Health Programme for drug prevention (Grant #SPC 2002376 and Grant #SPC 2005312).
  This questionnaire collects information, knowledge and opinions on substance use, with emphasis on alcohol, tobacco and drugs use. It also gather information about tobacco, alcohol, marijuana and other drugs use; and assess risk and protective factors. It consists of 45 questions. In the Chilean validation, all subscales had an acceptable internal reliability (omega > 0.65).
SURPS | One month
  The Substance Use Risk Profile Scale, is a self-reported questionnaire that gather information about anxiety sensitivity, hopelessness, sensation seeking, and impulsivity. These four sub scales have been associated as risk factors for drug use among adolescents. the internal reliability for each subscale is: anxiety sensitivity (alpha=0.65), hopelessness (alpha=0.76), sensation seeking (alpha=0.62), and impulsivity (alpha=0.61).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gaete, MD PhD, Principal Investigator — Universidad de los Andes, Chile
Locations (1):
- Universidad de los Andes, Santiago, Chile

REFERENCES:
- [Result] Faggiano F, Galanti MR, Bohrn K, Burkhart G, Vigna-Taglianti F, Cuomo L, Fabiani L, Panella M, Perez T, Siliquini R, van der Kreeft P, Vassara M, Wiborg G; EU-Dap Study Group. The effectiveness of a school-based substance abuse prevention program: EU-Dap cluster randomised controlled trial. Prev Med. 2008 Nov;47(5):537-43. doi: 10.1016/j.ypmed.2008.06.018. Epub 2008 Jul 9. PMID 18657569
- [Result] Faggiano F, Vigna-Taglianti F, Burkhart G, Bohrn K, Cuomo L, Gregori D, Panella M, Scatigna M, Siliquini R, Varona L, van der Kreeft P, Vassara M, Wiborg G, Galanti MR; EU-Dap Study Group. The effectiveness of a school-based substance abuse prevention program: 18-month follow-up of the EU-Dap cluster randomized controlled trial. Drug Alcohol Depend. 2010 Apr 1;108(1-2):56-64. doi: 10.1016/j.drugalcdep.2009.11.018. Epub 2010 Jan 18. PMID 20080363
- [Result] Vigna-Taglianti FD, Galanti MR, Burkhart G, Caria MP, Vadrucci S, Faggiano F; EU-Dap Study Group. "Unplugged," a European school-based program for substance use prevention among adolescents: overview of results from the EU-Dap trial. New Dir Youth Dev. 2014 Spring;2014(141):67-82, 11-2. doi: 10.1002/yd.20087. PMID 24753279
- [Result] Faggiano F, Richardson C, Bohrn K, Galanti MR; EU-Dap Study Group. A cluster randomized controlled trial of school-based prevention of tobacco, alcohol and drug use: the EU-Dap design and study population. Prev Med. 2007 Feb;44(2):170-3. doi: 10.1016/j.ypmed.2006.09.010. Epub 2006 Nov 3. PMID 17084887
- [Result] Prado MC, Schneider DR, Sanudo A, Pereira AP, Horr JF, Sanchez ZM. Transcultural Adaptation of Questionnaire to Evaluate Drug Use Among Students: The Use of the EU-Dap European Questionnaire in Brazil. Subst Use Misuse. 2016;51(4):449-58. doi: 10.3109/10826084.2015.1117108. Epub 2016 Feb 19. PMID 26894657
- [Result] Sanchez ZM, Valente JY, Sanudo A, Pereira APD, Cruz JI, Schneider D, Andreoni S. The #Tamojunto Drug Prevention Program in Brazilian Schools: a Randomized Controlled Trial. Prev Sci. 2017 Oct;18(7):772-782. doi: 10.1007/s11121-017-0770-8. PMID 28361199
- [Result] Newton NC, Barrett EL, Castellanos-Ryan N, Kelly E, Champion KE, Stapinski L, Conrod PJ, Slade T, Nair N, Teesson M. The validity of the Substance Use Risk Profile Scale (SURPS) among Australian adolescents. Addict Behav. 2016 Feb;53:23-30. doi: 10.1016/j.addbeh.2015.09.015. Epub 2015 Sep 25. PMID 26441044
- [Result] Woicik PA, Stewart SH, Pihl RO, Conrod PJ. The Substance Use Risk Profile Scale: a scale measuring traits linked to reinforcement-specific substance use profiles. Addict Behav. 2009 Dec;34(12):1042-55. doi: 10.1016/j.addbeh.2009.07.001. Epub 2009 Jul 8. PMID 19683400
- [Derived] Salgado G, Gaete J, Gana S, Valenzuela D, Araya R. Acceptability, feasibility and fidelity of the culturally adapted version of Unplugged ("Yo Se Lo Que Quiero"), a substance use preventive program among adolescents in Chile: a pilot randomized controlled study. BMC Public Health. 2024 Jul 29;24(1):2026. doi: 10.1186/s12889-024-19499-2. PMID 39075465